CLINICAL TRIAL: NCT06653348
Title: De-Escalation of Dual Antiplatelet Therapy With Ticagrelor and Aspirin in Non-disabling Non-cardioembolic Ischemic Stroke or High Risk TIA Patients: A Randomized, Outcome Assessor Blind, Controlled Trial
Brief Title: Ticagrelor Based De-Escalation of Dual Antiplatelet Therapy in Ischemic Stroke
Acronym: DEDAPT-TICA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Athena Sharifi Razavi, Dr. Athena Sharifi Razavi, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23439; mazmus (Other Grant/Funding Number: mazandaran university of medical sciences)
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: ischemic stroke; non-cardioembolic; non-disabling; TIA; Ticagrelor; de-escalation; dual antiplatelet therapy
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient | interventions — Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study designed to be blind to the outcome assessors, meaning that the neurologist evaluating the patients' outcomes was unaware of the treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Intervention group will be treat with ASA 325 mg stat and ticagrelor 180 mg stat, then ASA 80 mg daily and ticagrelor 90 mg BID for 30 days. Then ticagrelor 60 mg BID and ASA 80 mg daily until the end of month 6.
  Interventions: Drug: Ticagrelor 60 + Aspirin
- comparator (Active Comparator): Comparator group will be treat with ASA 325 mg stat and ticagrelor 180 mg stat, then ASA 80 mg daily and ticagrelor 90 mg BID for 30 days. Then ASA 80 mg daily until the end of month 6.
  Interventions: Drug: Ticagrelor 90 + aspirin

INTERVENTIONS:
Drug: Ticagrelor 60 + Aspirin — Ticagrelor 90 mg BID plus ASA 80 mg daily for 1 month and then ticagrelor 60 mg BID plus ASA 80 mg daily until the end of month 6.
  Arms: intervention
Drug: Ticagrelor 90 + aspirin — ticagrelor 90 mg BID plus ASA 80 mg daily for 1 month.
  Arms: comparator

SUMMARY:
This is a randomized, controlled, outcome assessor blind, parallel group design pilot study on 100 patient with diagnosis of ischemic stroke admitted in Bou-Ali Sina Hospital, Sari,Iran.The aim of study is to compare the efficacy of 90 mg ticagrelor BID plus aspirin for 1 month and 60 mg ticagrelor BID plus aspirin for 6 months in reduce of non-disabling non-cardioembolic ischemic stroke or high risk TIA recurrence during first 12 months.

DETAILED DESCRIPTION:
This is a randomized, controlled, parallel, outcome assessor blind, feasibility study. The aim of study is assess the efficacy of ticagrelor de-escalation in reduce of non-disabling non-cardioembolic ischemic stroke or high risk TIA recurrence during first 12 months after primary event. 100 patient with diagnosis of ischemic stroke admitted in Bou-Ali Sina Hospital, Sari, Iran will be randomized to intervention or control group by using 4 block randomization method. Inclusion criteria is : age>40, signing inform consent, recent ischemic stroke within 24 h, diagnosed by brain CT or MRI mild stroke with NIHSS =<8 and no evidence of large infarct in brain imaging.,high risk TIA with ABCD >4, no cardioembolic source such as low E/F, MS, AF ,... no specific etiology such as dissection, vasculitis, ... no carotid stenosis > 50 % in side of involvement. Exclusion criteria is :history of hypersensitivity to consumptive drug any indication for anticoagulant therapy acute phase treatment with intravenous thrombolysis or thrombectomy any contraindication for consumptive drug history of intracranial hemorrhage history of GI bleeding during past 6 m candidate for endarterectomy history of coagulopathy active hemorrhagic diathesis during randomization. Patients in control group will be treat with standard ischemic stroke regiment including ASA 325 mg stat and ticagrelor 180 mg stat, then ASA 80 mg and ticagrelor 90 mg BID for 1 month. Then single antiplatelet therapy with ASA will be continue. Intervention group will be treat with ASA 325 mg stat and ticagrelor 180 mg stat, then ASA 80 mg daily and ticagrelor 90 mg BID for 1 month. And, Ticagrelor 60 mg BID plus ASA 80 mg daily until the end of month 6. Then single antiplatelet therapy with ASA will be continue. Four fallow up visit plan by a neurologist or neurology resident on month 1, 3, 6 and 12.Clinical data including NIHSS score, MRS score and other data will record on case report form. Stroke recurrence or cardiovsacular event is efficacy end point. Major bleeding according to STIH criteria is study safety end point. Primary outcome is ischemic stroke recurrence during first 12 months after first event documented by new lesion on brain CT or MRI. Secondary outcome is major hemorrhagic events, stroke recurrence during first 6 months and any cardiovascular event during first 12 month.

ELIGIBILITY:
Inclusion Criteria:

* signing inform consent,
* recent ischemic stroke within 24 h,
* diagnosed by brain CT or MRI mild stroke with NIHSS =<8 and no evidence of large infarct in brain imaging
* high risk TIA with ABCD >4,
* no cardioembolic source such as low E/F, MS, AF ,...
* no specific etiology such as dissection, vasculitis, ...
* no carotid stenosis > 50 % in side of involvement

Exclusion Criteria:

* history of hypersensitivity to consumptive drug
* any indication for anticoagulant therapy
* acute phase treatment with intravenous thrombolysis or thrombectomy
* any contraindication for consumptive drug
* history of intracranial hemorrhage
* history of GI bleeding during past 6 m
* candidate for endarterectomy
* history of coagulopathy
* active hemorrhagic diathesis during randomization

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
ischemic stroke recurrence | 12 months
  recording new event based on new lesion on brain CT scan or MRI

SECONDARY OUTCOMES:
Major hemorrhagic event | during first 180 days
  Major bleeds were defined according to the International Society of Thrombosis and Hemostasis (ISTH)

CONTACTS AND LOCATIONS:
Locations (1):
- Mazandaran province, Sari,Iran, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: Undecided